CLINICAL TRIAL: NCT02960412
Title: Randomized Controlled Trial Evaluating Effect of Furosemide on Confirmation of Ureteral Patency During Routine Cystoscopy
Brief Title: Effect of Furosemide on Confirmation of Ureteral Patency During Routine Cystoscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: Pro00026976
Record Dates: First submitted 2016-11-07; First posted 2016-11-09 (Estimated); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Cystoscopy
MeSH Terms: interventions — Furosemide; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- furosemide (Experimental): furosemide 10mg (1mL) IV push for one dose
  Interventions: Drug: furosemide
- placebo (Placebo Comparator): normal saline 1mL IV push for one dose
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: furosemide — 10mg lasix given intraoperatively
  Other Names: Lasix
  Arms: furosemide
Drug: Normal Saline — Normal saline given intraoperatively as placebo
  Arms: placebo

SUMMARY:
This study evaluates if administration of IV furosemide leads to expedited confirmation of ureteral patency when compared to placebo (IV saline) in routine cystoscopy performed after urogynecologic surgery.

DETAILED DESCRIPTION:
Cystoscopy is performed routinely after urogynecologic surgery to ensure there was no injury to the urinary tract (urethra, bladder, or ureters). In order to confirm that no damage occurred to the ureters, a jet of urine must be visualized from each ureteral opening.

The time it takes to confirm this ureteral patency is variable and some sources suggest using furosemide to decrease the time it takes to see these jets. This study will evaluate what effect, if any, this medicine has on time to confirming ureteral patency.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing any urogynecologic surgery
* No allergy or contraindication to receiving furosemide
* Normal Creatinine/glomerular filtration rate

Exclusion Criteria:

* Unable to consent, including if non English speaking
* Allergy or contraindication to receiving furosemide
* Intraoperative injury to the lower urinary tract

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
time to ureteral patency | intra-operative
  time to confirmation of ureteral patency in seconds

SECONDARY OUTCOMES:
adverse effects from furosemide administration | immediately post operative (1-3 days post operatively)

CONTACTS AND LOCATIONS:
Locations (1):
- Tampa General Hospital, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Patton S, Tanner JP, Prieto I, Jackson E, Greene K, Bassaly R, Wyman AM. Furosemide Use and Time to Confirmation of Ureteral Patency During Intraoperative Cystoscopy: A Randomized Controlled Trial. Obstet Gynecol. 2019 Apr;133(4):669-674. doi: 10.1097/AOG.0000000000003155. PMID 30870291